CLINICAL TRIAL: NCT06216119
Title: Intrarenal Venous Flow Change During Fluid Removal in Critically Ill Patients: A Prospective Exploratory Study
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: SI929/2023
Record Dates: First submitted 2023-12-19; First posted 2024-01-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness; Fluid Overload
Keywords: critical illness; intrarenal venous flow pattern; fluid removal; venous excess ultrasound score; Renal Doppler ultrasonography; lung ultrasound
MeSH Terms: conditions — Critical Illness; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This clinical trial aims to study intrarenal venous flow patterns change, VExUS score change, and LUS score change during fluid removal treatment in critically ill patients

DETAILED DESCRIPTION:
Background: In patients with heart failure, intrarenal venous flow patterns could change depending on the level of congestion and was strongly correlated with death from cardiovascular disease and unplanned hospitalization. However, the findings may differ in patients with sepsis in the intensive care unit. In this case, Intrarenal venous flow patterns were not associated with Central Venous Pressure but were associated with Acute Kidney Injury and death. This suggests that intrarenal venous flow patterns may serve as an indicator of renal congestion and could be a feasible bedside tool to predict various clinical implications. In addition, Point-of-care ultrasound (POCUS) techniques such as Venous Excess Ultrasound (VExUS) and Lung Ultrasound (LUS) provide non-invasive assessments of fluid status and venous congestion. This study evaluates changes in VExUS and LUS scores during fluid removal to predict clinical outcomes in critically ill patients.

Objective: We aimed to study intrarenal venous flow patterns change, VExUS score change, and LUS score change during fluid removal treatment in critically ill patients.

Methods:

* After enrollment, patients will undergo baseline Doppler ultrasonography to evaluate intrarenal venous flow patterns and LUS before the initiation of fluid removal through diuretic therapy or renal replacement therapy.
* After patients received fluid removal therapy, they will receive continuous ultrasonography monitoring within 24, 48, and 72 hours, along with data collection.

Researchers will collect data about

* intrarenal venous flow patterns change, Venous Excess Ultrasound (VExUS) score change, and LUS score change during fluid removal treatment
* establish a correlation between alterations in intrarenal flow patterns, VExUS score, and LUS score as well as other clinical data (Central venous pressure, Cumulative fluid balance) and clinical implications (Renal replacement therapy free day, Ventilator free day, length of Intensive care unit stay).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years old or older who will be admitted to the medical intensive care unit
2. Expected to be hospitalized in the intensive care unit for more than 120 hours.
3. The patient has stable vital signs without the need for vasoactive medications or rapid fluid resuscitation (at least 500 milliliters of colloid or 1000 milliliters of crystalloid via rapid intravenous infusion) for a minimum consecutive period of 12 hours. This includes cases where the patient receives norepinephrine at a rate not exceeding 0.1 micrograms per kilogram per minute and dobutamine at a rate not exceeding 10 micrograms per kilogram per minute, or when the patient can maintain a continuous reduction in vasoactive medications for a minimum consecutive period of 12 hours.
4. The patient does not exhibit signs suggestive of inadequate organ perfusion, such as mottling skin, a capillary refill time of more than 2 seconds when nailbeds are pressed and released, or cold extremities.
5. The patients require fluid removal through decisions made by attending staff or clinical guidelines, which may involve the administration of diuretics or Renal Replacement Therapy.

Exclusion Criteria:

1. Underlying chronic kidney disease (eGFR< 30) before enrollment
2. Chronic renal replacement therapy (RRT) before enrollment such as on intermittent hemodialysis, peritoneal dialysis
3. Decompensated cirrhosis with portal hypertension
4. Inferior vena cava, portal vein, hepatic, renal vein thrombosis
5. Ureteral obstruction
6. Intraabdominal hypertension (Intraabdominal pressure > 12 mmHg)
7. Previous allergic or anaphylactic to diuretic
8. Pregnant women
9. Transplanted kidney, transplanted liver
10. Patients with do-not-resuscitate (DNR) orders or decisions to withhold life-sustaining treatments
11. Patients or their legally authorized representatives (LAR), who decline participation in the study or are unable to provide informed consent before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18 years old or older who will be admitted to the medical intensive care unit and require fluid removal therapy
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-01-23 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
intrarenal venous flow patterns change during fluid removal treatment in critically ill patients. | 72 hours after Fluid removal therapy
  intrarenal venous flow patterns change measured by ultrasonography

SECONDARY OUTCOMES:
VExUS score change following fluid removal treatment in critically ill patients. | 72 hours after Fluid removal therapy
  VExUS score change measured by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Ranistha Ratanarat, MD, Principal Investigator — Division of Critical Care, Department of Medicine, Siriraj Hospital, Mahidol University; Apatsara Saokaew, MD, Study Director — Division of Critical Care, Department of Medicine, Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All Individual participant data that underlie results in a publication of this study (after deidentification)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All IPD will become available starting briefly following a publication of the study with no end date.
Access Criteria: Investigators whose proposed use of the data has been approved by institutional review board or ethical committee.

REFERENCES:
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Hoste EA, Maitland K, Brudney CS, Mehta R, Vincent JL, Yates D, Kellum JA, Mythen MG, Shaw AD; ADQI XII Investigators Group. Four phases of intravenous fluid therapy: a conceptual model. Br J Anaesth. 2014 Nov;113(5):740-7. doi: 10.1093/bja/aeu300. Epub 2014 Sep 9. PMID 25204700
- [Background] Zhang L, Chen Z, Diao Y, Yang Y, Fu P. Associations of fluid overload with mortality and kidney recovery in patients with acute kidney injury: A systematic review and meta-analysis. J Crit Care. 2015 Aug;30(4):860.e7-13. doi: 10.1016/j.jcrc.2015.03.025. Epub 2015 Apr 9. PMID 25979272
- [Background] Vaara ST, Pettila V, Kaukonen KM, Bendel S, Korhonen AM, Bellomo R, Reinikainen M; Finnish Acute Kidney Injury Study Group. The attributable mortality of acute kidney injury: a sequentially matched analysis*. Crit Care Med. 2014 Apr;42(4):878-85. doi: 10.1097/CCM.0000000000000045. PMID 24201174
- [Background] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385
- [Background] Claure-Del Granado R, Mehta RL. Fluid overload in the ICU: evaluation and management. BMC Nephrol. 2016 Aug 2;17(1):109. doi: 10.1186/s12882-016-0323-6. PMID 27484681
- [Background] Malbrain MLNG, Van Regenmortel N, Saugel B, De Tavernier B, Van Gaal PJ, Joannes-Boyau O, Teboul JL, Rice TW, Mythen M, Monnet X. Principles of fluid management and stewardship in septic shock: it is time to consider the four D's and the four phases of fluid therapy. Ann Intensive Care. 2018 May 22;8(1):66. doi: 10.1186/s13613-018-0402-x. PMID 29789983
- [Background] Koratala A, Ronco C, Kazory A. Diagnosis of Fluid Overload: From Conventional to Contemporary Concepts. Cardiorenal Med. 2022;12(4):141-154. doi: 10.1159/000526902. Epub 2022 Sep 12. PMID 36096121
- [Background] Beaubien-Souligny W, Rola P, Haycock K, Bouchard J, Lamarche Y, Spiegel R, Denault AY. Quantifying systemic congestion with Point-Of-Care ultrasound: development of the venous excess ultrasound grading system. Ultrasound J. 2020 Apr 9;12(1):16. doi: 10.1186/s13089-020-00163-w. PMID 32270297
- [Background] Iida N, Seo Y, Sai S, Machino-Ohtsuka T, Yamamoto M, Ishizu T, Kawakami Y, Aonuma K. Clinical Implications of Intrarenal Hemodynamic Evaluation by Doppler Ultrasonography in Heart Failure. JACC Heart Fail. 2016 Aug;4(8):674-82. doi: 10.1016/j.jchf.2016.03.016. Epub 2016 May 11. PMID 27179835
- [Background] Yamamoto M, Seo Y, Iida N, Ishizu T, Yamada Y, Nakatsukasa T, Nakagawa D, Kawamatsu N, Sato K, Machino-Ohtsuka T, Aonuma K, Ohte N, Ieda M. Prognostic Impact of Changes in Intrarenal Venous Flow Pattern in Patients With Heart Failure. J Card Fail. 2021 Jan;27(1):20-28. doi: 10.1016/j.cardfail.2020.06.016. Epub 2020 Jul 9. PMID 32652246
- [Background] Ter Maaten JM, Dauw J, Martens P, Somers F, Damman K, Metalidis C, Nijst P, Dupont M, Mullens W. The Effect of Decongestion on Intrarenal Venous Flow Patterns in Patients With Acute Heart Failure. J Card Fail. 2021 Jan;27(1):29-34. doi: 10.1016/j.cardfail.2020.09.003. Epub 2020 Sep 11. PMID 32927066
- [Background] Fujii K, Nakayama I, Izawa J, Iida N, Seo Y, Yamamoto M, Uenishi N, Terasawa T, Iwata M. Association between intrarenal venous flow from Doppler ultrasonography and acute kidney injury in patients with sepsis in critical care: a prospective, exploratory observational study. Crit Care. 2023 Jul 10;27(1):278. doi: 10.1186/s13054-023-04557-9. PMID 37430356
- [Background] Fan J, Upadhye S, Worster A. Understanding receiver operating characteristic (ROC) curves. CJEM. 2006 Jan;8(1):19-20. doi: 10.1017/s1481803500013336. No abstract available. PMID 17175625
- [Background] Macedo E, Bouchard J, Soroko SH, Chertow GM, Himmelfarb J, Ikizler TA, Paganini EP, Mehta RL; Program to Improve Care in Acute Renal Disease Study. Fluid accumulation, recognition and staging of acute kidney injury in critically-ill patients. Crit Care. 2010;14(3):R82. doi: 10.1186/cc9004. Epub 2010 May 6. PMID 20459609
- [Background] Vaara ST, Korhonen AM, Kaukonen KM, Nisula S, Inkinen O, Hoppu S, Laurila JJ, Mildh L, Reinikainen M, Lund V, Parviainen I, Pettila V; FINNAKI Study Group. Fluid overload is associated with an increased risk for 90-day mortality in critically ill patients with renal replacement therapy: data from the prospective FINNAKI study. Crit Care. 2012 Oct 17;16(5):R197. doi: 10.1186/cc11682. PMID 23075459
- [Derived] Maluangnon C, Saokaew A, Rojwatcharapibarn S, Ratanarat R. Intrarenal venous flow patterns and their association with successful fluid removal in critically ill patients: a prospective observational exploratory study. Ultrasound J. 2025 Oct 6;17(1):44. doi: 10.1186/s13089-025-00447-z. PMID 41051454